CLINICAL TRIAL: NCT01970930
Title: Treatment Strategies for Myeloproliferative Neoplasms by Targeting the Tumor Suppressor P53
Brief Title: Tissue Banking Study - Polycythemia Vera or Essential Thrombocythemia (PV & ET) Patients
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-0481
Record Dates: First submitted 2013-08-20; First posted 2013-10-28 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
Keywords: Tissue banking
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CD34+ cells isolated from the peripheral blood Splenic CD34+ cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PV or ET: subject who has polycythemia vera or essential thrombocythemia
  Interventions: Procedure: Blood specimen

INTERVENTIONS:
Procedure: Blood specimen — 4 green top tube 40 cc of blood draw

SUMMARY:
The purpose of the study is to isolate and characterize stem cells of patients with Polycythemia Vera (PV) and Essential Thrombocythemia (ET) to find out why these cells are not working the way they should be and why they seem to be sensitive to regulatory factors in the blood, such as clotting.

DETAILED DESCRIPTION:
Specific Aim 1: Assess the effects of RG7112 on MPN HSC/HPC p53 levels and study how it affects MPN stem cell function.

Specific Aim 2. Assess the effects of a combination of low doses of IFNα and RG7112 on MPN HSC/HPC.

ELIGIBILITY:
Inclusion Criteria:

* polycythemia vera or essential thrombocythemia
* agree to give blood for study

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have polycythemia vera or essential thrombocythemia
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Stem cell function | at one time study visit
  Assess the effects of RG7112 on MPN HSC/HPC p53 levels and study how it affects MPN stem cell function.

SECONDARY OUTCOMES:
CD34+ cells assays | at one time study visit
  Assess the effects of a combination of low doses of IFNα and RG7112 on MPN HSC/HPC. After treatment with RG7112 and IFNα at the various doses, p53, MDM2, MDMX, phosphor-p38, and phosphor-STAT1 levels in MPN CD34+ cells will be measured using monoclonal antibody staining and flow cytometric and immunofluorescence analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hoffman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States